CLINICAL TRIAL: NCT06778252
Title: UrbanHEAT: Pilot of Prospective Observational Study of Health Behaviors, Outcomes, and Disparities in Individually Experienced Temperature Across an Urban Community
Brief Title: UrbanHEAT: Health Behaviors, Outcomes, and Disparities in Individually Experienced Temperature Across an Urban Community
Status: Withdrawn | Type: Observational
Why Stopped: Departure of key research team members.
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Other Study IDs: 10002097; 002097-MD
Record Dates: First submitted 2025-01-15; First posted 2025-01-16 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Temperature
Keywords: Physical Activity; Observational Study; Sleep; Climate Change; Cardiometabolic Risk Behaviors and Outcomes; Stress/mental well-being; Neighborhoods; TEMPERATURE
MeSH Terms: conditions — Motor Activity; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Volunteers: Healthy Volunteers with home address in Washington, DC.

SUMMARY:
We are conducting a research study to learn about how individuals living in Washington, DC perceive and experience temperature.

Participation in this study will include:

2 remote visits over the phone and/or computer (these will each last about1.5 to 2 hours)

* During the remote visits, you will be asked to respond to a series of surveys, so that we can learn about your life, behaviors, and health

  2 weeks of data collection where you will be asked to:
* Wear monitoring devices

  * These will collect information on your location and physical activity
  * We will ask you to wear the monitors on a belt around your waist all day every day during these 2 weeks of data collection.
  * All of the monitors will be sent to you in the mail.
* Leave a temperature tracker near where you sleep to measure the temperature of your environment.
* Use a phone app

  * We will also send you questions through the phone app that will ask about your stress level, sleep duration, sleep quality, and how you feel about the current temperature.

Risks of participating in this study are minimal. They include the inconvenience of wearing the monitors and the possibility of a breach of your confidentiality. We are collecting personal information about you and the location monitor will collect information about where you spend your time. We will take every precaution in order to safeguard the data that you provide, including limiting who has access to it, storing it safely, and removing the capacity to identify you individually, as much as possible.

You will receive no immediate benefits from participating in this study. We hope what we learn will help us to develop policies and programs to help keep urban populations safe during increasingly warm summer temperatures.

You are eligible for this study if you are 18 years of age or older, live in Washington, DC, can read and write in English, and have access to a smartphone that you can use for the 2 week data collection period....

DETAILED DESCRIPTION:
Study Description:

This pilot study will test measures for cardiometabolic behaviors and outcomes (e.g., physical activity, sedentary behavior, stress, sleep quality, sleep quantity) and individually experienced temperature with intensive longitudinal data collected via wearable devices and smart phone-based ecological momentary assessment. The primary hypothesis is that there are associations between individually experienced temperature and the identified behaviors and outcomes.

Objectives:

Primary:

To explore within and between-person associations between individually experienced temperature and cardiometabolic risk behaviors and outcomes.

Secondary:

Aim 1: Explore disparities in individually experienced temperature based on race, ethnicity, socioeconomic factors, sex, and age.

Aim 2: Explore multilevel determinants of individually experienced temperature: neighborhood environment (residential and activity space), home, workplace, and preferences

Endpoints:

Primary:

* Physical Activity
* Sedentary behavior
* Stress/mental well-being
* Sleep quantity
* Sleep quality

Secondary:

* Daily mean individually experienced temperature
* Daily maximum individually experienced temperature
* Daily degree minutes above threshold
* Longest daily exposure period

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Ability of subject to understand and the willingness to sign a written informed consent document.
* Aged at least 18 years.
* Ability to read and write in English. This is justified by the novelty of the survey instruments (e.g., momentary thermal comfort conducted in an ecological momentary assessment context).
* Home address in Washington, DC
* Availability of a smart phone on which Metricwire Ecological Momentary Assessment software can be downloaded and used during the 14-day data collection period.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Requirement of hospitalization at enrollment.
* Inability to consent.
* Unwillingness to comply with study procedures.

Ages: 18 Years to 115 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults 18 and over with home addresses located within Washington, DC.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-07-22 (Actual); Primary Completion 2025-07-29 (Actual); Study Completion 2025-07-29 (Actual)

PRIMARY OUTCOMES:
Physical Activity | 2 weeks
  Daily/Weekly Minutes MVPA (Moderate to Vigorous Physical Activity) as measured via waist-worn acceleromter
Sedentary Behavior | 2 weeks
  Daily/Weekly Minutes Sedentary Behavior as measured via waist-worn accelerometer
Stress/mental Well-being | 2 weeks
  Momentary/Daily Mean/Weekly Mean score on ecological momentary assessment random prompt questions derived from PSS-4 stress survey
Sleep Quantity | 2 weeks
  Daily/Weekly Mean Hours Sleep collected via daily ecological momentary assessment morning prompt
Sleep Quality | 2 weeks
  Daily/Weekly Mean Score derived from PSQI sleep survey collected via daily ecological momentary assessment morning prompt

SECONDARY OUTCOMES:
Daily mean individually experienced temperature | 2 weeks
  average of all daily minute-epoch individual environmental temperature measures collected via iButton Hygrochron aggregated to (1) 24-hour days, (2) daylight only days, and (3) nighttime only days
Daily maximum individually experienced temperature | 2 weeks
  highest measured minute-epoch individual environmental temperature collected via iButton Hygrochron for (1) 24-hour days, (2) daylight only days, and (3) nighttime only days
Daily degree minutes above threshold | 2 weeks
  minutesXdegrees exceeding test thresholds ranging from 80F-105F collected via iButton Hygrochron for (1) 24-hour days, (2) daylight only days, and (3) nighttime only days
Longest daily exposure period | 2 weeks
  minutes of longest daily period exceeding test thresholds ranging from 80F-105F collected via iButton Hygrochron for (1) 24-hour days, (2) daylight only days, and (3) nighttime only days

CONTACTS AND LOCATIONS:
Overall Officials: Kelly K Jones, Principal Investigator — National Institute on Minority Health and Health Disparities (NIMHD)
Locations (1):
- National Institute on Minority Health and Health Disparities, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Aggregated, non-identifiable data will be submitted to a data repository as required by policy.

REFERENCES:
- [Background] Beyer KMM, Szabo A, Hoormann K, Stolley M. Time spent outdoors, activity levels, and chronic disease among American adults. J Behav Med. 2018 Aug;41(4):494-503. doi: 10.1007/s10865-018-9911-1. Epub 2018 Jan 30. PMID 29383535
- [Background] Tran Trong T, Riera F, Rinaldi K, Briki W, Hue O. Ingestion of a cold temperature/menthol beverage increases outdoor exercise performance in a hot, humid environment. PLoS One. 2015 Apr 9;10(4):e0123815. doi: 10.1371/journal.pone.0123815. eCollection 2015. PMID 25856401
- [Background] Kuras ER, Richardson MB, Calkins MM, Ebi KL, Hess JJ, Kintziger KW, Jagger MA, Middel A, Scott AA, Spector JT, Uejio CK, Vanos JK, Zaitchik BF, Gohlke JM, Hondula DM. Opportunities and Challenges for Personal Heat Exposure Research. Environ Health Perspect. 2017 Aug 1;125(8):085001. doi: 10.1289/EHP556. PMID 28796630
- [Background] McGregor GR, Vanos JK. Heat: a primer for public health researchers. Public Health. 2018 Aug;161:138-146. doi: 10.1016/j.puhe.2017.11.005. Epub 2017 Dec 28. PMID 29290376
- [Background] Song X, Wang S, Hu Y, Yue M, Zhang T, Liu Y, Tian J, Shang K. Impact of ambient temperature on morbidity and mortality: An overview of reviews. Sci Total Environ. 2017 May 15;586:241-254. doi: 10.1016/j.scitotenv.2017.01.212. Epub 2017 Feb 7. PMID 28187945
- [Background] Waugh DW, He Z, Zaitchik B, Peng RD, Diette GB, Hansel NN, Matsui EC, Breysse PN, Breysse DH, Koehler K, Williams D, McCormack MC. Indoor heat exposure in Baltimore: does outdoor temperature matter? Int J Biometeorol. 2021 Apr;65(4):479-488. doi: 10.1007/s00484-020-02036-2. Epub 2020 Oct 21. PMID 33089367
- [Background] White-Newsome JL, Sanchez BN, Jolliet O, Zhang Z, Parker EA, Dvonch JT, O'Neill MS. Climate change and health: indoor heat exposure in vulnerable populations. Environ Res. 2012 Jan;112:20-7. doi: 10.1016/j.envres.2011.10.008. Epub 2011 Nov 8. PMID 22071034
- [Background] Xiang J, Bi P, Pisaniello D, Hansen A. Health impacts of workplace heat exposure: an epidemiological review. Ind Health. 2014;52(2):91-101. doi: 10.2486/indhealth.2012-0145. Epub 2013 Dec 21. PMID 24366537
- [Background] Zuurbier M, van Loenhout JAF, le Grand A, Greven F, Duijm F, Hoek G. Street temperature and building characteristics as determinants of indoor heat exposure. Sci Total Environ. 2021 Apr 20;766:144376. doi: 10.1016/j.scitotenv.2020.144376. Epub 2020 Dec 26. PMID 33421789